CLINICAL TRIAL: NCT00436579
Title: A Dose Escalation Study of Sorafenib (BAY 43-9006, NSC 724772) in Nomotensive Patients With Advanced Malignancies
Brief Title: Sorafenib in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00221; NCI-2009-00221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-15002A; CDR0000528261; 15002A (Other: University of Chicago); 7768 (Other: CTEP); U01CA069852 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Sorafenib

ARMS (3):
- Arm I (higher-dose enzyme inhibitor therapy) (Experimental): Patients receive higher-dose oral sorafenib tosylate twice daily on days 15-36.
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Procedure: assessment of therapy complications; Other: laboratory biomarker analysis
- Arm II (standard-dose enzyme inhibitor therapy) (Active Comparator): Patients receive standard-dose oral sorafenib tosylate three times daily on days 15-36.
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Procedure: assessment of therapy complications; Other: laboratory biomarker analysis
- Arm III (standard-dose enzyme inhibitor therapy) (Active Comparator): Patients receive standard-dose oral sorafenib tosylate twice daily on days 15-36. (closed to accrual as of 4/29/2009)
  Interventions: Drug: sorafenib tosylate; Other: pharmacological study; Procedure: assessment of therapy complications; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study
  Other Names: pharmacological studies
Procedure: assessment of therapy complications — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial is studying the side effects, such as high blood pressure, and best dose of sorafenib in treating patients with advanced solid tumors. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether increasing the dose of sorafenib tosylate increases the plasma steady-state concentration in patients with advanced solid tumors.

II. Determine whether increasing the dose of this drug affects blood pressure in these patients.

SECONDARY OBJECTIVES:

I. Determine whether the variability in blood pressure elevation is due to pharmacokinetic or pharmacodynamic variability.

II. Compare the toxicity and differences in pharmacokinetics of delivering a higher dose of this drug per day (using two different schedules) vs delivering the currently recommended dose of this drug.

III. Investigate mechanisms of sorafenib tosylate-induced hypophosphatemia with serial measurements of phosphate metabolism (no longer assessed as of 4/29/2009) in these patients, detailed baseline measurements in all patients, and detailed evaluations of patients developing grade 3 or greater hypophosphatemia.

IV. Detect subclinical effects of this drug on measures of thyroid function. V. Identify biomarkers predicting the categorization of patient response.

OUTLINE: This is a randomized, dose-escalation study.

Patients receive oral sorafenib tosylate twice daily on days 1-7 and once on day 8. Patients not experiencing at least one grade 2 or higher toxicity during the initial sorafenib treatment are randomized to 1 of 3 dose-escalated treatment arms.

ARM I: Patients receive higher-dose oral sorafenib tosylate twice daily on days 15-36.

ARM II: Patients receive standard-dose oral sorafenib tosylate three times daily on days 15-36.

ARM III: (closed to accrual as of 4/29/2009) Patients receive standard-dose oral sorafenib tosylate twice daily on days 15-36.

In all arms, treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo ambulatory blood pressure monitoring at baseline, on days 7, 14, and 21, and at 6 and 12 months. Blood samples are collected periodically throughout study and evaluated for pharmacokinetic studies, thyroid function, serum markers, and phosphate metabolism*. CT perfusion imaging is performed at baseline, week 6, week 12, and then every 8-12 weeks thereafter.

NOTE: * Phosphate metabolism no longer assessed as of 4/29/2009.

After completion of study treatment, patients are followed every 4 weeks for 1 year and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant solid tumor

  * Refractory disease for which curative or palliative measures have failed or for which there is no known superior treatment
  * No colorectal cancer or melanoma
* Measurable OR nonmeasurable disease
* Normotensive (blood pressure [BP] ≤ 140/90 mm Hg) meeting 1 of the following criteria:

  * No more than 2 attempted measurement sessions for which the documented mean systolic BP is ≤ 140 mm Hg and the diastolic BP is ≤ 90 mm Hg
  * At least 30 attempted measurement sessions for which the documented mean systolic BP is ≤ 135 mm HG and the diastolic BP is ≤ 85 mm Hg
* Brain metastases allowed provided the following criteria are met:

  * Stable neurologic status for ≥ 2 weeks after completion of definitive local therapy (surgery or radiotherapy)
  * No neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Age ≥ 14 years OR weight ≥ 45 kilograms (pediatric patients)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if there is liver involvement)
* Creatinine ≤ 1.5 times ULN
* No New York Heart Association class II-IV congestive heart failure
* No unstable angina (anginal symptoms at rest) or new-onset angina (began within the past 3 months)
* No myocardial infarction within the past 6 months
* No ventricular arrhythmias requiring anti-arrhythmic therapy
* No thrombotic or embolic events, such as symptomatic pulmonary embolus or any cerebrovascular accident (including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage/bleeding event > grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event > grade 3 within the past 4 weeks
* No evidence or history of bleeding diathesis or coagulopathy
* No serious nonhealing wound, ulcer, or bone fracture
* No ongoing or active infection > grade 2
* No psychiatric illness or social situation that would limit compliance with study requirements
* No allergy to sorafenib tosylate or excipients
* No unstable condition that would jeopardize the safety of the patient and/or her/his compliance with the study
* No significant traumatic injury within the past 4 weeks
* No condition that would impair the patient's ability to swallow whole pills or capacity to absorb oral medications
* No seizure disorder requiring steroids or anticonvulsant therapy
* No other concurrent illness
* Recovered from prior therapy
* Prior vascular endothelial growth factor (VEGF) pathway inhibitor (e.g., bevacizumab, sunitinib malate, axitinib) allowed provided the following criteria are met:

  * The patient's best response as measured by RECIST criteria was not progressive disease
  * If the most recent agent was a small molecule reversible inhibitor (e.g., sunitinib malate, cediranib, or axitinib), the patient must not have taken a dose of the agent within 2 weeks of the baseline blood pressure session and 3 weeks of starting sorafenib tosylate
  * If the most recent agent was bevacizumab or VEGF trap the patient must not have received the most recent dose within 5 weeks of the baseline blood pressure session and 6 weeks of starting sorafenib tosylate AND no grade 3 bleeding, cardiovascular, skin, or thyroid toxicities on one of these previous therapies
* More than 2 weeks since prior and no concurrent radiotherapy
* At least 3 weeks since prior and no concurrent chronic epoetin alfa (or congeners)
* More than 3 weeks since prior immunotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior major surgery or open biopsy
* At least 3 weeks since prior uncharacterized herbal agents or nutritional supplements
* More than 12 weeks since prior radioimmunotherapy
* No prior sorafenib tosylate
* No prior organ allograft or allogeneic bone marrow or peripheral blood stem cell transplantation

  * Patients with a history of autologous transplant and normal bone marrow function are eligible
* No prior cyclosporine, Hypericum perforatum (St. John's wort), or rifampin
* No other concurrent investigational agents
* No other concurrent antineoplastic therapy, including chemotherapy, except androgen-ablating agents (for patients with prior prostate cancer)
* No concurrent hematopoietic growth factors
* No concurrent combination antiretroviral therapy for HIV-positive or chronic hepatitis B-positive patients
* No concurrent hormonal therapy except steroids for adrenal insufficiency or hormones for nondisease-related conditions (e.g., insulin for diabetes)

  * Steroids for autoimmune cytopenia allowed provided dose has been stable for 3 weeks
* No anticipated need for other antineoplastic therapy within the next 4 weeks

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in BP | From baseline to day 21
  BP will first be calculated for each subject as BP after 1 week of treatment minus BP before that treatment dose. Then, for each randomized group separately, the BP changes in the two study phases will be compared using paired t-tests.

SECONDARY OUTCOMES:
Association between steady state trough levels of sorafenib and BP | Days 8 and 22
  Spearman correlation coefficients (since the distribution of sorafenib plasma trough levels is not normal and the relationship may be non-linear) will be calculated and scatter plots will be produced separately for each phase of the study. The association between differences in trough levels at the two different doses and changes in BP due to dose escalation will be tested in a similar manner. comparisons of BP changes and drug plasma levels between the three randomized treatment arms will be analyzed by analysis of variance (ANOVA) followed by Tukey's allowance for multiple comparisons.
Toxicity rates in the two high dose groups | Every 2 weeks, assessed up to 1 year
  Toxicity rates will be summarized by type, grade, and attribution and compared using chi-squared tests or Fisher exact tests, as appropriate.
Effect of sorafenib dose/exposure on thyroid function | From baseline up to 50 days
  Analysis of variance for repeated measures with one between groups factor (sorafenib dose) and one within subjects factor (time) will be used on serum parathyroid hormone (PTH).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States